CLINICAL TRIAL: NCT03415230
Title: Effect of Therapeutic Massage on Sleep Quality and Stress Levels in Women With Breast Cancer: A Randomized Control Trial
Brief Title: Effect of Therapeutic Massage on Sleep Quality and Stress Levels in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Collaborators: Cyprus Anticancer Society (Unknown)
Responsible Party: Principal Investigator, Dr. Andreas Charalambous, Associate Professor, Cyprus University of Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC-TMSQ-2018
Record Dates: First submitted 2018-01-09; First posted 2018-01-30 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Sleep Disturbance; Anxiety
MeSH Terms: conditions — Parasomnias; Anxiety Disorders | interventions — Massage

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: therapeutic massage vs sham massage
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic massage (Experimental): Women will undertake sessions of therapeutic massage
  Interventions: Other: Therapeutic massage
- Sham massage (Sham Comparator): Women will undertake sessions of sham massage
  Interventions: Other: Sham massage

INTERVENTIONS:
Other: Therapeutic massage — Massage therapy involves the administration of combinations of specific physical manipulations applied in a systematic way, with varying intensity, direction, rate, and rhythm, to the soft tissues of the body.
  Arms: Therapeutic massage
Other: Sham massage — Sham massage involves only light touch massage in a non systematic way
  Arms: Sham massage

SUMMARY:
This is a randomized control trial to test the effectiveness of therapeutic massage on the sleep quality and the stress levels in women that have completed their treatment for breast cancer.

DETAILED DESCRIPTION:
The period following the completion of treatment for breast cancer (but also for any other type of cancer as well) is once that is accompanied by an increased uncertainty. This can often trigger increased anxiety levels and sleep disturbances. This trial tests the effectiveness of therapeutic massage as a non pharmaceutical intervention that can increase the management of stress and sleep disturbances during this period of time.

ELIGIBILITY:
Inclusion Criteria:

* Women that completed their treatment
* women experiencing insomnia
* women experiencing anxiety
* women that speak and understand Greek

Exclusion Criteria:

* allergy to essential oils
* use of anticoagulants
* presence of edema
* presence of Varicose veins

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with Breast Cancer
Enrollment: 40 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
Sleep Disturbances (insomnia) | Change from baseline total score at 4 weeks
  Athens insomnia scale (The AIS is a self-assessment psychometric instrument designed for quantifying sleep difficulty based on the ICD-10 criteria. It consists of eight items: the first five pertain to sleep induction, awakenings during the night, final awakening, total sleep duration, and sleep quality; while the last three refer to well-being, functioning capacity, and sleepiness during the day). Each item of the AIS can be rated 0-3, (with 0 corresponding to no problem at all and 3 to very serious problem); thus, the total score ranges from 0 (absence of any sleep-related problem) to 24 (the most severe degree of insomnia).

SECONDARY OUTCOMES:
Anxiety | Change from baseline total score at 4 weeks
  Hamilton Anxiety Rating Scale (HAM-A). The scale consists of 14 items. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Charalambous, PhD, Principal Investigator — Cyprus University of Technology
Locations (1):
- Oncology Centre, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided
Demographic information can be shared